CLINICAL TRIAL: NCT00717561
Title: A National, Prospective, Randomized, Open Label Study to Assess the Efficacy and Safety of IV/PO Moxifloxacin vs IV Ceftriaxone + IV Azithromycin Followed by PO Amoxicilline/Clavulanate and PO Clarithromycin in Subjects With Community-acquired Pneumonia
Brief Title: A Study to Assess the Efficacy and Safety of IV/PO Moxifloxacin in Subjects With Community-acquired Pneumonia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12669; 2007-001320-12 (EudraCT Number)
Record Dates: First submitted 2008-07-16; First posted 2008-07-17 (Estimated); Last update posted 2014-11-04 (Estimated); Status verified 2014-10

CONDITIONS: Pneumonia
Keywords: CAP; Community-acquired pneumonia
MeSH Terms: conditions — Pneumonia; Community-Acquired Pneumonia | interventions — Moxifloxacin; Ceftriaxone; Azithromycin; Amoxicillin; Clavulanic Acid; Clarithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Avelox (Moxifloxacin, BAY12-8039)
- Arm 2 (Active Comparator)
  Interventions: Drug: Ceftriaxone; Azithromycin; Amoxicilline/clavulanate; Clarithromycin

INTERVENTIONS:
Drug: Avelox (Moxifloxacin, BAY12-8039) — IV therapy: every 24 hours, patients will be administered a 400 mg moxifloxacin infusion over 60 minutes. Oral therapy: patients will be administered a single moxifloxacin 400 mg tablet, every 24 hours
  Arms: Arm 1
Drug: Ceftriaxone; Azithromycin; Amoxicilline/clavulanate; Clarithromycin — IV therapy: every 24 hours patients will be administered a 2 g ceftriaxone infusion over 30 minutes. Following the infusion with ceftriaxone, patients will be administered a 500 mg azithromycin infusion over 180 minutes.Oral therapy: every 8 hours patients will be administered a 1000 mg amoxicillin/clavulanic acid tablet. Every 12 hours patients will be administered a 500 mg clarithromycin tablet.
  Arms: Arm 2

SUMMARY:
The purpose of this study is to assess if a therapy with oral and intravenous moxifloxacin is as effective as a therapy with intravenous ceftriaxone + intravenous azithromycin followed by oral amoxicilline/clavulanate and oral clarithromycin in the treatment of community-acquired pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized non-ICU patients (age, >= 18 years)
* Clinical signs and symptoms of CAP, with PSI score IV or V
* Radiologically confirmed evidence of a new and/or progressive infiltrate(s)
* Requirement for initial parenteral therapy
* At least 2 of the following conditions:

  * Productive or non productive cough with or without purulent or mucosus or mucopurulent sputum
  * Dyspnea and/or tachypnea (respiratory rate of > 20 breaths/min)
  * Rigors and/or chills
  * Pleuritic chest pain
  * Auscultatory findings of rales and/or crackles on pulmonary examination and/or evidence of pulmonary consolidation
  * Fever (an oral temperature of >= 38 °C, a rectal temperature of >= 39 °C, or a tympanic temperature of >= 38.5 °C) or hypothermia (rectal or core temperature of < 35 °C), and a WBC count of >= 10,000 cells/mm3 or >= 15% immature neutrophils bands; regardless of peripheral WBC count) or leukopenia (total WBC count of < 4500 cells/mm3)
* Written informed consent

Exclusion Criteria:

* PSI Class I-III and V with need for ICU admission
* Hospitalization for > 48 hours before developing pneumonia, or discharge from hospital < 30 days prior. Note: patients currently residing in residential long-term facilities can be enrolled in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-02; Primary Completion 2009-05 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Clinical response 20 days after completion of study treatment (Test-of-Cure visit) | 20 days after last dose of study drug (TOC Visit)

SECONDARY OUTCOMES:
Clinical and bacteriological response on the day of switch from IV to oral therapy | Day of switch from IV to oral therapy
Clinical and bacteriological response on treatment Day 3-5 (if the day of switch is different from Day 3, 4 or 5) | Day 3-5
Bacteriological response at TOC | 20 days after last dose of study drug
Clinical and bacteriological response at the end of treatment | Day 7-14 after first dose of study drug
Mortality attributable to pneumonia at the Test-of-Cure visit | 20 days after last dose of study drug

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (20):
- Italy (20):
  - Lungro, Cosenza
  - San Cesario di Lecce, Lecce
  - Fossombrone, Pesaro e Urbino
  - Pregiato Di Cava Dei Tirreni, Salerno
  - Vittorio Veneto, Treviso
  - Ascoli Piceno
  - Benevento
  - Brescia
  - Catania
  - Chieti
  - Foggia
  - Lucca
  - Macerata
  - Messina
  - Milan
  - Palermo
  - Roma
  - Sassari
  - Torino
  - Udine

REFERENCES:
- See also: Click here and search for information provided by EMA — http://www.clinicaltrialsregister.eu